CLINICAL TRIAL: NCT01332500
Title: Treximet ™ Pharmacy Budget Impact Model Database Validation Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111208
Record Dates: First submitted 2011-03-21; First posted 2011-04-11 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Migraine Disorders
Keywords: Triptans; Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; sumatriptan-naproxen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- adult migraineurs with/without aura: Adult migraine patients >18-65 years who have initiated treatment for migraine with Treximet ™ or other orally administered triptan.
  Interventions: Drug: Sumatriptan/Naproxen combination; Drug: other oral triptans

INTERVENTIONS:
Drug: Sumatriptan/Naproxen combination — Sumatriptan and Naproxen Sodium
  Other Names: Treximet (TM)
Drug: other oral triptans — almotriptan, eletriptan, frovatriptan, naratriptan, rizatriptan, sumatriptan, zolmitriptan

SUMMARY:
The purpose of this retrospective claims database study was to compare the change in migraine-related prescription (i.e. NSAIDs, Opioids, Ergots) utilization among migraine suffers following initiation of Treximet ™ (sumatriptan/naproxen) compared with subjects initiating treatment with other orally available triptans. The study was used to validate the migraine-related prescription utilization patterns predicted by the Treximet ™ Budget Impact Model.

The SourceLx dataset from the family of Wolters Kluwer databases was used for this analysis. The database contains 30% of prescription claims filled in the United States (US), approximately 160 million patient lives. The data has broad representative coverage at both the geographic and payment levels.

ELIGIBILITY:
Inclusion Criteria:

* At least one prescription claim for either Treximet ™ or orally administered triptan
* at least 18 years of age at index Rx date
* at least one prescription claim for any medication in the pre- and post-index period (proxy for continuous enrollment)

Exclusion Criteria:

* Subjects receiving nasal sumatriptan at any time
* Subjects over 65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject data from a claims database having at least one pharmacy claim for Treximet ™ or an orally administered triptan during the study period.
Sampling Method: Probability Sample
Enrollment: 61737 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Naïve - Sumatriptan/Naproxen Sodium: Participants having at least one pharmacy claim for sumatriptan/naproxen sodium or an orally administered triptan during January 1, 2007 to November 30, 2009 (study period) were selected as the target population. The index date was defined as the fill date of the first chronologically occurring sumatriptan-naproxen sodium/oral triptan prescription during the enrollment period (January 1, 2009 to May 31, 2009). Participants belonged to this arm if their first prescription was for sumatriptan/naproxen sodium. Sumatriptan/naproxen sodium users were matched to oral triptan users on propensity scores based on baseline characteristics.
- Naïve - Oral Triptan: Participants having at least one pharmacy claim for sumatriptan/naproxen sodium or an orally administered triptan during January 1, 2007 to November 30, 2009 (study period) were selected as the target population. The index date was defined as the fill date of the first chronologically occurring sumatriptan-naproxen sodium/oral triptan prescription during the enrollment period (January 1, 2009 to May 31, 2009). Participants belonged to this arm if their first prescription was for an oral triptan.
- Switch - Sumatriptan/Naproxen Sodium: Participants having at least one pharmacy claim for sumatriptan/naproxen sodium or an orally administered triptan during January 1, 2007 to November 30, 2009 (study period) were selected as the target population. The index date was defined as the date of first switch to sumatriptan/naproxen sodium or an oral triptan prescription during the enrollment period (January 1, 2009 to May 31, 2009). Participants belonged to this arm if they received oral triptan as their first triptan medication and then switched to sumatriptan/naproxen sodium in the enrollment period. Sumatriptan/naproxen sodium users were matched to oral triptan users on propensity scores based on baseline characteristics.
- Switch - Oral Triptan: Participants having at least one pharmacy claim for sumatriptan/naproxen sodium or an orally administered triptan during January 1, 2007 to November 30, 2009 (study period) was selected as the target population. The index date was defined as the date of first switch to sumatriptan/naproxen sodium or an oral triptan prescription during the enrollment period (January 1, 2009 to May 31, 2009). Participants belonged to this arm if they received oral triptan as their first triptan medication and then switched to a different oral triptan in the enrollment period. Sumatriptan/naproxen sodium users were matched to oral triptan users on propensity scores based on baseline characteristics.
Period: Overall Study
Arm/Group | Naïve - Sumatriptan/Naproxen Sodium | Naïve - Oral Triptan | Switch - Sumatriptan/Naproxen Sodium | Switch - Oral Triptan
Started | 13257 | 39771 | 2903 | 5806
Completed | 13257 | 39771 | 2903 | 5806
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Naïve - Oral Triptan: Participants having at least one pharmacy claim for sumatriptan/naproxen sodium or an orally administered triptan during January 1, 2007 to November 30, 2009 (study period) were selected as the target population. The index date was defined as the fill date of the first chronologically occurring sumatriptan-naproxen sodium/oral triptan prescription during the enrollment period (January 1, 2009 to May 31, 2009). Participants belonged to this arm if their first prescription was for an oral triptan.
  Sumatriptan/naproxen sodium users were matched to oral triptan users on propensity scores based on baseline characteristics.
- Total: Total of all reporting groups
Arm/Group | Naïve - Sumatriptan/Naproxen Sodium | Naïve - Oral Triptan | Switch - Sumatriptan/Naproxen Sodium | Switch - Oral Triptan | Total
Number analyzed (Participants) | 13257 | 39771 | 2903 | 5806 | 61737
Age, Customized [Number; unit: Participants]
  18-30 years old | 2889 | 8867 | 464 | 1026 | 13246
  31-40 years old | 3425 | 10172 | 669 | 1251 | 15517
  41-50 years old | 3700 | 10887 | 943 | 1763 | 17293
  51-60 years old | 2315 | 6993 | 610 | 1263 | 11181
  61-70 years old | 758 | 2368 | 191 | 428 | 3745
  >70 years old | 170 | 484 | 26 | 75 | 755
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11108 | 33371 | 2525 | 5078 | 52082
  Male | 2149 | 6400 | 378 | 728 | 9655

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Triptan Tablets Per Participant in 6-month Follow-up Period: Treatment-naïve Analysis
Description: The mean number of tablets per participant was computed using prescription fills dispensed in the 6-month follow-up period. "Other" represents acetaminophen (APAP)/isometheptene/dichlorphenazone and APAP/isometheptene/caffeine, for example. The number of tablets dispensed was obtained from the "quantity dispensed field" in the claims data. Triptan tablets were classified as index and non-index medication (if a different oral triptan was filled from that of the index medication); only oral triptans were considered (i.e., excluded injectable triptans).
Time Frame: 6-months from the index date (from January 1, 2009 to May 31, 2009; the index date was defined as the first date of oral triptan/sumatriptan-naproxen sodium prescription)
Population: The SourceLx dataset from the family of Wolters Kluwer databases was used for this study. The database contains 30% of prescription claims filled in the United States, corresponding to approximately 160 million lives.
Measure: Mean (Standard Deviation); unit: tablets per participant
Arm/Group | Naïve - Sumatriptan/Naproxen Sodium | Naïve - Oral Triptan
Number analyzed (Participants) | 13257 | 39771
tablets per participant
  Triptans | 17.7 (16.3) | 18.4 (18.2)
  Non-steroidal anti-inflammatory drugs | 19.2 (57.1) | 21.5 (64.9)
  Opioids | 75.8 (219.0) | 80.1 (235.8)
  Ergots | 0.1 (3.6) | 0.1 (2.4)
  Other | 1.5 (17.0) | 1.4 (13.9)
Statistical Analysis 1: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Triptan tablets
Statistical Analysis 2: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Non-steroidal anti-inflammatory drug tablets
Statistical Analysis 3: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.005, paired t-test 2-sided — Opioid tablets
Statistical Analysis 4: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.336, paired t-test 2-sided — Ergot tablets
Statistical Analysis 5: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.162, paired t-test 2-sided — Other tablets

2. Primary Outcome: Mean Health Plan Cost Per Participant for Migraine-related Medications in 6-month Follow-up Period: Treatment-naïve Analysis
Description: Health plan cost was defined as the pharmacy costs. Pharmacy costs were computed corresponding to the use of triptans, non-steroidal anti-inflammatory drugs, opioids, and other migraine therapy tablets (ergots and others). Pharmacy costs were calculated as the mean of the total costs of the five drug categories.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Naïve - Sumatriptan/Naproxen Sodium | Naïve - Oral Triptan
Number analyzed (Participants) | 13257 | 39771
United States dollars
  Triptans | 284 (366.1) | 333 (393.7)
  Non-steroidal anti-inflammatory drugs | 9 (62.3) | 9 (62.5)
  Opioids | 38 (609.7) | 43 (477.6)
  Ergots | 2 (33.1) | 2 (51.2)
  Other | 0 (5.1) | 0 (4.8)
  Total | 332 (732.1) | 387 (645.4)
Statistical Analysis 1: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Triptan health plan costs
Statistical Analysis 2: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.349, paired t-test 2-sided — Non-steroidal anti-inflammatory drug health plan costs
Statistical Analysis 3: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.208, paired t-test 2-sided — Opioid health plan costs
Statistical Analysis 4: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.239, paired t-test 2-sided — Ergot health plan costs
Statistical Analysis 5: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.583, paired t-test 2-sided — Other health plan costs
Statistical Analysis 6: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Total heath plan costs

3. Primary Outcome: Mean Total Cost (Health Plan Plus Participant Copay Costs) Per Participant for Migraine-related Medications in 6-month Follow-up Period: Treatment-naïve Analysis
Description: Mean Total Cost was defined as the pharmacy cost plus the participant copay. Pharmacy costs were computed corresponding to the use of triptans, non-steroidal anti-inflammatory drugs, opioids, and other migraine therapy tablets (ergots and others). Pharmacy cost plus participant copay was calculated as the mean of the total costs (pharmacy cost plus participant copay) of the five drug categories.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Naïve - Sumatriptan/Naproxen Sodium | Naïve - Oral Triptan
Number analyzed (Participants) | 13257 | 39771
United States dollars
  Triptans | 349 (396.4) | 397 (418.9)
  Non-steroidal anti-inflammatory drugs | 11 (69.8) | 12 (72.5)
  Opioids | 49 (621.0) | 54 (509.5)
  Ergots | 2 (36.6) | 2 (55.5)
  Other | 1 (8.6) | 1 (7.2)
  Total | 412 (757.7) | 466 (687.7)
Statistical Analysis 1: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Triptan health plus copay costs
Statistical Analysis 2: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.177, paired t-test 2-sided — Non-steroidal, anti-inflammatory drug health plus copay costs
Statistical Analysis 3: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.173, paired t-test 2-sided — Opioid health plus copay costs
Statistical Analysis 4: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.191, paired t-test 2-sided — Ergot health plus copay costs
Statistical Analysis 5: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p = 0.254, paired t-test 2-sided — Other health plus copay costs
Statistical Analysis 6: Comparison: Naïve - Sumatriptan/Naproxen Sodium vs Naïve - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Total health plus copay costs

4. Primary Outcome: Mean Number of Triptan Tablets Per Participant in 6-month Follow-up Period: Treatment-switch Analysis
Description: The mean number of tablets per participant was computed using prescription fills dispensed in the 6-month follow-up period. "Other" represents APAP/isometheptene/dichlorphenazone and APAP/isometheptene/caffeine, for example. The number of tablets dispensed was obtained from the "quantity dispensed field" in the claims data. Triptan tablets were classified as index and non-index medication (if a different oral triptan was filled from that of the index medication); only oral triptans were considered (i.e., excluded injectable triptans).
Time Frame: 6-months from the index date (from January 1, 2009 to May 31, 2009; index date was defined as the first switch date to oral triptan/sumatriptan-naproxen sodium prescription)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: tablets per participant
Arm/Group | Switch - Sumatriptan/Naproxen Sodium | Switch - Oral Triptan
Number analyzed (Participants) | 2903 | 5806
tablets per participant
  Triptans | 24.4 (20.7) | 24.4 (20.2)
  Non-steroidal anti-inflammatory drugs | 20.9 (62.5) | 22.9 (70.9)
  Opioids | 88.4 (254.7) | 87.4 (255.7)
  Ergots | 0.0 (1.6) | 0.1 (3.7)
  Other | 1.4 (14.9) | 1.3 (12.1)
Statistical Analysis 1: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.866, paired t-test 2-sided — Triptan tablets
Statistical Analysis 2: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.094, paired t-test 2-sided — Non-steroidal anti-inflammatory drug tablets
Statistical Analysis 3: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.832, paired t-test 2-sided — Opioid tablets
Statistical Analysis 4: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.392, paired t-test 2-sided — Ergot tablets
Statistical Analysis 5: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.752, paired t-test 2-sided — Other tablets

5. Primary Outcome: Mean Health Plan Cost Per Participant for Migraine-related Medications in 6-month Follow-up Period: Treatment-switch Analysis
Description: Health Pan Cost was defined as the pharmacy costs. Pharmacy costs were computed corresponding to the use of triptans, non-steroidal anti-inflammatory drugs, opioids, and other migraine therapy tablets (ergots and others). Pharmacy costs were calculated as the mean of the total costs of the five drug categories.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Switch - Sumatriptan/Naproxen Sodium | Switch - Oral Triptan
Number analyzed (Participants) | 2903 | 5806
United States dollars
  Triptans | 375 (374.5) | 425 (413.3)
  Non-steroidal anti-inflammatory drugs | 8 (52.5) | 10 (67.2)
  Opioids | 47 (317.8) | 51 (522.9)
  Ergots | 3 (48.9) | 3 (50.1)
  Other | 0 (6.7) | 0 (3.9)
  Total | 433 (507.4) | 490 (695.8)
Statistical Analysis 1: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Triptan health plan costs
Statistical Analysis 2: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.054, paired t-test 2-sided — Non-steroidal anti-inflammatory drug health plan costs
Statistical Analysis 3: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.590, paired t-test 2-sided — Opioid health plan costs
Statistical Analysis 4: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.382, paired t-test 2-sided — Ergot health plan costs
Statistical Analysis 5: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.343, paired t-test 2-sided — Other health plan costs
Statistical Analysis 6: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Total health plan costs

6. Primary Outcome: Mean Total Cost (Health Plan Plus Participant Copay Costs) Per Participant for Migraine-related Medications in 6-month Follow-up Period: Treatment-switch Analysis
Description: Mean Total Cost was defined as the pharmacy cost plus the participant copay. Pharmacy costs were computed corresponding to the use of triptans, non-steroidal anti-inflammatory drugs, opioids, and other migraine therapy tablets (ergots and others). .Pharmacy cost plus participant copay was calculated as the mean of the total costs (pharmacy cost plus participant copay) of the five drug categories.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States dollars
Arm/Group | Switch - Sumatriptan/Naproxen Sodium | Switch - Oral Triptan
Number analyzed (Participants) | 2903 | 5806
United States dollars
  Triptans | 462 (413.3) | 496 (439.9)
  Non-steroidal anti-inflammatory drugs | 12 (62.3) | 13 (76.7)
  Opioids | 61 (360.2) | 62 (547.4)
  Ergots | 3 (51.9) | 4 (54.4)
  Other | 1 (8.5) | 1 (6.1)
  Total | 537 (564.2) | 576 (736.2)
Statistical Analysis 1: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p < 0.001, paired t-test 2-sided — Triptan health plus copay costs
Statistical Analysis 2: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.146, paired t-test 2-sided — Non-steroidal anti-inflammatory drug health plus copay costs
Statistical Analysis 3: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.826, paired t-test 2-sided — Opioid health plus copay costs
Statistical Analysis 4: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.354, paired t-test 2-sided — Ergot health plus copay costs
Statistical Analysis 5: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.514, paired t-test 2-sided — Other health plus copay costs
Statistical Analysis 6: Comparison: Switch - Sumatriptan/Naproxen Sodium vs Switch - Oral Triptan; Test type: Superiority or Other; p = 0.001, paired t-test 2-sided — Total health plus copay costs

ADVERSE EVENTS:
Description: This study was a retrospective, observational cohort study with the primary purpose of assessing migraine-specific pharmacy utilization and costs associated with initiating/switching to sumatriptan/naproxen sodium compared to other oral triptans. Therefore, adverse event information was not captured.
Arm/Group | Naïve - Sumatriptan/Naproxen Sodium | Naïve - Oral Triptan | Switch - Sumatriptan/Naproxen Sodium | Switch - Oral Triptan
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.